CLINICAL TRIAL: NCT01673230
Title: Hemodynamic Indices Predictive of a Beneficial Response to Fluid Expansion in Case of Hemodynamic Failure After Cardiac Surgery With Altered Preoperative Ejection Fraction (LVEF≤45%): Sensibility and Specificity of Respiratory Variations of Pulse Pressure (∆PP), Photoplethysmography (∆POP), Perfusion Index (PVI), Before and After Fluid Expansion.
Brief Title: Hemodynamic Indices Predictive of a Beneficial Response to Fluid Expansion in Case of Hemodynamic Failure After Cardiac Surgery With Altered Preoperative Ejection Fraction (LVEF≤45%)
Acronym: ALTERVOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2012-A00364-39; LOC/12-01 (Other: Rennes University Hospital (Direction of Clinical Research))
Record Dates: First submitted 2012-08-22; First posted 2012-08-27 (Estimated); Last update posted 2019-12-27 (Actual); Status verified 2016-03

CONDITIONS: Ventricular Dysfunction
MeSH Terms: conditions — Ventricular Dysfunction | interventions — Cardiac Surgical Procedures

ARMS (1):
- Ventricular dysfunction (Other): cardiac surgery for ventricular dysfunction
  Interventions: Procedure: cardiac surgery for ventricular dysfunction

INTERVENTIONS:
Procedure: cardiac surgery for ventricular dysfunction — For each included patient during the immediate post operative period, hemodynamic variables will be recorded (continuous arterial pressure, ECG, photoplethysmographic curve, CVP, wedge pressure, respiratory pressure), at rest (proclive 45°), during fluid expansion (physiological saline).

SUMMARY:
Low Cardiac Output Syndrome occurs frequently after cardiac surgery, especially when pre-operative LVEF is altered (LVEF≤45%). The correction of hemodynamic failure requires adapted treatments: fluid expansion and/or inotropic or vasoactive drugs. Predictive indices of a response to fluid challenge may allow an earlier hemodynamic optimization, which has not been showed until now when LVEF is altered.

ELIGIBILITY:
Inclusion Criteria:

* patients >18 years old in the immediate post-operative period after cardiac surgery
* ASA 1 - 3
* Pre-operative LVEF≤45%
* Sedated with Ramsay score: 6
* Mechanically ventilated with tidal volume at 8ml/kg, PEEP at 0mmHg, I/Eat 0,5
* With hemodynamic failure: SAP≤90mmHg and/or inotropic or vasoactive drug started in the operating room and/or clinical sign of shock and/or CI ≤2,3l/min/m2
* Affiliation to Health Insurance
* Consent form signed

Exclusion Criteria:

* Cardiac arrhythmia: frequent atrial or ventricular extra systoles, atrial fibrillation
* Intracardiac shunt
* Weight less than 50 kg
* History of central nervous system illness
* Pulmonary oedema (clinical and/or radiological and/or wedge pressure>18mmHg)
* Right ventricular failure suspected (CVP> wedge pressure) or diagnosed (trans thoracic and/or transesophageal echocardiography)
* Acute kidney injury with oligoanuria
* Severe post operative bleeding (chest tubes volume of >200ml/h for 3 hours or more)
* Severe hypoxia (PaO2/FIO2< 100)
* Administrative control (patient under guardianship or curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Measure of ∆PP, ∆POP, PVI and Cardiac index (CI) | 2 hours
  To assess the sensibility and specificity of ∆PP, ∆POP, PVI, after fluid expansion in case of hemodynamic failure in the immediate post-operative period after cardiac surgery, when pre-operative LVEF is altered.

SECONDARY OUTCOMES:
Measure of Systolic, diastolic and mean arterial pressure (SAP, DAP, MAP), Central venous pressure (CVP) and wedge pressure. | 2 hours
  Secondary objectives :
  * Early optimization of hemodynamics after cardiac surgery,
  * To determine optimal threshold for ∆PP, ∆POP and PVI,
  * To compare dynamic (∆PP, ∆POP and PVI) with static (central venous pressure: CVP, wedge pressure) indices

CONTACTS AND LOCATIONS:
Overall Officials: patrick guinet, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France